CLINICAL TRIAL: NCT06385691
Title: Evaluation of the Efficacy of the myDIET Software Tool in the Nutritional Management of Patients With Localized and Resectable Gastric or Esogastric Junction Cancer.
Brief Title: Study Evaluating the Efficacy of the myDIET Software Tool in the Nutritional Management of Patients With Localized and Resectable Gastric or Esogastric Junction Cancer.
Acronym: MyDIET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ET22-145
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer; Oesogastric Junction Cancer
Keywords: denutrition; software tool; physical activity; postoperative chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm Phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of myDIET tool for nutritional management (Experimental): Patients will be followed up at regular intervals during neoadjuvant chemotherapy, perioperatively and up to 6 months after the date of surgery (after completion of postoperative chemotherapy).
  Interventions: Other: myDIET software tool

INTERVENTIONS:
Other: myDIET software tool — The tool is based on self-questionnaires completed by the patient. They are mainly filled in using visual analogue scales (from 0-10) or grades of symptoms/toxicities (Grades 0 to 4), based on the CTCAE V5. These scales will cover the following themes: food intake, weight changes, digestive symptoms, taste disorders, pain and fatigue. The system will be able to monitor data changes and the response given will be adapted according to the severity of symptoms:
  * No signs of seriousness: general prevention or treatment documents/advice: toxicity management, nutritional advices targeted on symptoms, on digestive problems, on appropriate physical activity.
  * Presence of signs of seriousness: action to be taken and alert to the coordinating nurse, oncologist or dietician.
  In case of an alert, the coordinating nurse will call the patient back and either manage the symptom, schedule a nutritional consultation to initiate nutritional management, or refer the patient to the oncologist.

SUMMARY:
This is a prospective, single-center, single-arm Phase II study evaluating the efficacy of the myDIET software tool in the nutritional management of patients with localized and resectable esogastric junction cancer.

DETAILED DESCRIPTION:
Gastric cancer is the 3rd leading cause of cancer mortality worldwide, with a 5-year survival rate of less than 30%. In localised gastric cancer (GC) or cancer of the oesogastric junction (OGJ), the standard treatment consists of gastrectomy and peri-operative FLOT-based chemotherapy (5FU, Leucovorin, Oxaliplatin, Taxotere). However, up to 51% of patients have post-operative complications, and only 60% can benefit from post-operative chemotherapy (at least one course) initiated within 12 weeks of surgery, while 46% receive the full theoretical regimen.

An incomplete adjuvant chemotherapy regimen drastically reduces post-operative prognosis. Undernutrition and sarcopenia increase the occurrence of post-operative complications, length of stay and post-operative readmissions. Undernutrition is an independent risk factor for failure and/or incomplete adjuvant chemotherapy, with an impact on progression-free survival and overall survival. There is a high prevalence of undernutrition in patients with GC/OGJ, estimated at 53-60%, and the proportion of undernourished patients increases significantly postoperatively compared with preoperatively.

Preoperative nutrition and physical activity in sarcopenic patients has been shown to reduce postoperative complications. Early multimodal management, combining nutrition, adapted physical activity and neoadjuvant chemotherapy, is therefore recommended and essential in the perioperative situation. To optimise the nutritional management of patients with operable gastric or oesogastric junction cancer, the CLB teams have developed a computer interface (MyDIET) linked to the myCLB patient portal. This provides semi-personalised monitoring based on self-questionnaires designed to assess and educate patients or their carers about nutritional issues from the outset of oncology treatment, and to prevent the onset or worsening of undernutrition.

For this reason, the sponsor proposes an exploratory study to assess the efficacy of the myDIET digital tool in increasing the proportion of patients with localised CG/OGJ initially treated with neo-adjuvant chemotherapy and who undergo surgery and are able to receive adjuvant chemotherapy within 8 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older at date of signing informed consent to participate;
* Histologically proven diagnosis of gastric adenocarcinoma or OGJ;
* Localized, resectable disease;
* Patient treated with perioperative Oxaliplatin-based chemotherapy,
* Performance status (ECOG): 0-2;
* Membership of a social security scheme;
* Signed informed consent to participate.

Exclusion Criteria:

* Other associated solid cancer or haemopathy;
* Presence of severe comorbidity (Charlson index < 9)
* Presence of unbalanced dysthyroidism (TSH not within laboratory norm at inclusion, usually between 0.4 and 4 mUI/L);
* History of gastric, duodenal or esophageal surgery;
* Inability to comply with study requirements, including :

  * Impossibility for the patient or his/her caregiver to connect to myDIET;
  * Difficulty in understanding the written French language;
  * Psychological incapacity (e.g. excessive vulnerability, psychiatric disorder) or physical incapacity (e.g.

physical/motor disability);

* Patient under guardianship, curatorship or safeguard of justice;
* Patients already participating in a clinical trial or interventional study likely to interfere with the evaluation of the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients starting adjuvant chemotherapy within 2 months | 2 months after surgery
  proportion of patients for whom adjuvant chemotherapy could be initiated within 2 months after surgery

SECONDARY OUTCOMES:
Adherence to the tool | From inclusion and up to 6 months after surgery
  Percentage of completed questionnaires
Number of supportive care and emergency consultations initiated by the caregiver | From inclusion and up to 6 months after surgery
  Number of supportive care and emergency consultations initiated by the caregiver on the bases of questionnaires completed by patients
Proportion of patients with malnutrition | From inclusion and up to 6 months after surgery
  Proportion of patients with malnutrition defined according to the criteria of the French National Authority for Health
Evolution of body composition in L3 section (volumes) | From inclusion and up to 6 months after surgery
  Evolution of body composition based on body composition in L3 section on CT scan in volumes (cm2) at inclusion, after neoadjuvant chemotherapy and 6 months after surgery.
Evolution of body composition in L3 section (indexes) | From inclusion and up to 6 months after surgery
  Evolution of body composition based on body composition in L3 section on CT scan in indexes (cm2/m2) at inclusion, after neoadjuvant chemotherapy and 6 months after surgery.
Evolution of resting energy expenditure | From inclusion and up to 1 month after surgery
  Changes in resting energy expenditure (Kcal/day) will be measured at inclusion, at day 7 postoperatively, and at 1 month after surgery (before adjuvant chemotherapy) with the measurement of basal metabolic rate quantified by indirect calorimetry (Kcal/day)
Proportion of patient covering theoretical nutritional requirement >= 30kcal/kg/day | From inclusion and up to 6 months after surgery
  The proportion of patients with dietary intakes > or equal to 30kcal/kg/day will be quantified during the dietary consultation at inclusion, at day 7 after surgery, at 1 month after surgery and 6 months after surgery.
Comparison between theoretical nutritional requirement and measurement of basal metabolic rate using indirect calorimetry | From inclusion and up to 6 months after surgery
  Theoretical nutritional requirement and measurement of basal metabolic rate using indirect calorimetry (kcal/day) will be quantified during the dietary consultation at inclusion, at day 7 after surgery, at 1 month after surgery and 6 months after surgery.
Weight changes | From inclusion and up to 6 months after surgery
  Weight changes will be described by the weight in kg
Brachial circumference changes | From inclusion and up to 6 months after surgery
  Brachial circumference will be described in cm
Triceps skin fold changes | From inclusion and up to 6 months after surgery
  Triceps skin fold will be described in mm
Initiation time for post-operative chemotherapy | From surgery to date of post operative chemotherapy initiation assessed up to 6 months after surgery
  Initiation time for post-operative chemotherapy will be defined as the time in days between the date of surgery and the date of the first course of post operative chemotherapy
Proportion of patient with incomplete scheme of pre operative chemotherapy | From inclusion to surgery
  Proportion of patient with incomplete scheme of pre operative chemotherapy and their causes will be described
Proportion of patient with incomplete scheme of post operative chemotherapy | From surgery and up to 6 months after surgery
  Proportion of patient with incomplete scheme of post operative chemotherapy and their causes will be described
Proportion of patients with severe post operative complication | From surgery up to 6 months ater surgery
  Proportion of patients with severe post operative complication will be described according to the occurence of a grade > III complication according to Clavien Dindo classification
Tolerance to perioperative chemotherapy | From inclusion up to 6 months after surgery
  Tolerance to perioperative chemotherapy will be assessed with self-assessment using myDIET questionnaires based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5 classification.
  Grades range from 1 to 5 and refer to the severity of the adverse event. A higher grade means a worse outcome.
Changes in food intake | From inclusion up to 6 months after surgery
  Changes in food intake will be evaluated during chemotherapy and the postoperative period (myDIET follow-up questionnaires).
Changes in SEFI (Easy Food Intake Score) | From inclusion up to 6 months after surgery
  Changes in SEFI (Easy Food Intake Score) will be evaluated using visual scales (during chemotherapy and the postoperative period (myDIET follow-up questionnaires).
  SEFIs are assessed using visual scales ('analogue' or 'portions eaten'). With the visual analogue scale, the patients indicate the quantities they are currently eating using the cursor on the graduated scale from "nothing at all" = 0 to "as usual" = 10.
  With the visual portions eatenscale , patients can use the cursor to indicate the portions eaten at their last meal (lunch or dinner).
Measurement of quality of life | From inclusion and up to 6 months after surgery
  Quality of life will be assessed with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This 30-item questionnaire is completed by the patient and includes five multi-item functional scales (physical, role, cognitive, emotional and social); eight symptom scales (fatigue, pain, nausea and vomiting, dyspnoea, insomnia, loss of appetite and constipation); and a global health scale. The score for each item ranges from 1 (not at all) to 4 (very much).
Average lengh of hospital stay | At the time of surgery, an average of 3 months
  The average lengh of hospital stay during surgery will be described in terms of the number of days spent in hospital
Recurrence free survival (RFS) | From inclusion and up to the date of radiologically documented relapse or death from any cause, whichever came first, assessed up to 30 months
  Recurrence free survival (RFS) will be definied as the duration in days between the date of inclusion and the date of radiologically documented relapse or death from any cause
Overall survival (OS) | From inclusion and up to the date of death from any cause, assessed up to 30 months
  Overall survival (OS) will be defined as the time in days from date of the inclusion to the date of death from any cause
Adherence to the physical activity program | From inclusion and up to 6 months after surgery
  Adherence to the physical activity program will be described by the number of weekly session declared by the patient
Physical activity levels | From inclusion and up to 6 months after surgery
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (short version). The questions ask how much time the patient has spent being physically active over the last 7 days (duration of activity in minutes or hours, and number of days of activity in days).
Assessment of muscular function by the 6-min walk test | From inclusion and up to 6 months after surgery
  Assessment of muscular function will be assessed by the 6-min walk test (described in meters)
Assessment of muscular function by muscular strength | From inclusion and up to 6 months after surgery
  Assessment of muscular function will be assessed by muscular strength measured with hand grip dynamometer (described in kg)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Funk-Debleds, MD, Principal Investigator — Centre Léon Berard
Locations (1):
- Centre Léon Berard, Lyon, France